CLINICAL TRIAL: NCT03793075
Title: Immune-mediatory Response of Intravenous Ketamine Versus Propofol for Major Abdominal Surgeries: a Prospective Randomized Study
Brief Title: Ketamine Versus Propofol Effect on the Immune-mediatory Response for Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Abdelraouf Elsharkawy, Lecturer of anesthesia and surgical intensive care, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R/18.09.287
Record Dates: First submitted 2018-12-30; First posted 2019-01-04 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Major Abdominal Surgery
MeSH Terms: interventions — Ketamine; Propofol

STUDY DESIGN:
Intervention Model Description: Participating subject will be divided equally and randomly into two groups.The first group is propofol group while the second is the ketamine group
Who Masked: Participant, Care Provider
Masking Description: Double -blinded ( masking of both participant and care provider)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol group (P) (Placebo Comparator): The maintenance of anesthesia , patient will receive sevoflurane 1%-2.5% with intravenous infusion of propofol 17 mcg /kg/min and 0.5 mg/kg fentanyl will be given if the heart rate or mean blood pressure increased by 30 % or more from the basal readings
  Interventions: Drug: Propofol
- Ketamine group ((K) (Active Comparator): The maintenance of anesthesia , patient will receive sevoflurane 1%-2.5% with intravenous infusion of ketamine 5 mcg /kg/min and 0.5 mg/kg fentanyl will be given if the heart rate or mean blood pressure increased by 30 % or more from the basal readings
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — ketamine 5 mcg/kg/min will be used as intravenous anesthetic infusion
  Other Names: ketalar
  Arms: Ketamine group ((K)
Drug: Propofol — propofol 17 mcg /kg/min
  Other Names: diprivan
  Arms: Propofol group (P)

SUMMARY:
Host systemic responses to vigorous stimuli as trauma, surgical tissue injury, anesthesia and post-operative pain, leads to release a variety of pro-inflammatory cytokines including interleukin-1 (IL-1) and interleukin-6 (IL-6) mainly from monocytes and macrophages Thus, the rise of IL-6 is regarded as an early marker of tissue damage and its rise proportional to the degree of tissue damage .

It has been demonstrated that systemic responses to stress may be modified by the anesthetic technique used . Total intravenous anesthesia (TIVA) especially propofol based greatly suppresses the stress response induced by surgery when compared to inhalation by lowering cortisol levels.

Ketamine has the ability to modulate (modify) inflammation . Even the sub-anesthetic doses of ketamine in animal models were even provided to have an effect on the inflammatory response system in the central nervous system

DETAILED DESCRIPTION:
The release a variety of pro-inflammatory cytokines including tumor necrosis factor-α (TNF-α), interleukin-1 (IL-1) and interleukin-6 (IL-6) mainly from monocytes and macrophages due to surgical trauma or anesthesia .

IL-6 is constantly found in the peripheral blood and rapidly within few minutes unlike other pro inflammatory mediators. Thus, the rise of IL-6 is regarded as an early marker of tissue damage and IL-6 levels are proportional to the degree of tissue damage . The two major actions of IL-6 are having a key role in regulating stress responses by activating the hypothalamic-pituitary- adrenal (HPA) axis and synthesizing fibrinogen (which is necessary for the acute-phase response) serving as a growth factor for activated B-cells .

While appropriate inflammatory reactions are advantageous and essential for wound healing and host defense against microorganisms, excessive immune responses can be detrimental. The released mediators prompt systemic endocrine, immunological and metabolic responses result in increased pain sensitivity, altered metabolism, hyperthermia and greater secretion of liver acute phase proteins and stress hormones, so yields unstable patient's hemodynamic status

Propofol was documented to have an advantage in terms of inflammatory and immunomodulatory effects through significant effect on TNF-α, IL-6 and IL-10 release .

Ketamine has the ability to modulate (modify) inflammation and this is why it is recommended in patients with sepsis undergoing surgery . This may be possibly related with the variations in TNF-α and nuclear factor-κB expression . Even the sub-anesthetic doses of ketamine in animal models were even provided to have an effect on the inflammatory response system in the central nervous system which is involved in its therapeutic effect on depression (Yang-2 et al., 2013).

This study will be conducted to compare between the intravenous infusion of ketamine against the intravenous infusion of propofol during general anesthesia in patients undergoing major abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Elective major abdominal surgeries with median incision with right or left extension.
* ASA -physical status I -II
* aged from 18 till 70 years

Exclusion Criteria:

* body mass index more than 35 kg/m2,
* Patients having severe cardiovascular, respiratory, hepatic, renal, Endocrinol disorders, malignant
* Patients having chronic inflammatory diseases
* Patients received suppressant drugs in the 6 weeks before surgery.
* Any known allergy or any contraindications to anesthetic drugs;
* patient refusal,
* The usage of anti- emetic drug 24 hours before operation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-01-10 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Serum level of interleukin 6 (IL-6) | The time frame extend from 10 minutes before the induction of anesthesia till the first 24 hours postoperative
  picogram/milliliter using ELISA techniques .Five measurement points : before the induction of general anesthesia, 30 min after beginning infusion of the anesthetic agent , then 2h, 8h and 24 hours postoperative.
Serum level of interleukin IL-1β (IL-1β) | The time frame extend from 10 minutes before induction of anesthesia till the first 24 hours postoperative
  picogram/milliliter using ELSA techniques .Five measurement points : before the induction of general anesthesia, 30 min after beginning infusion of the anesthetic agent , then 2h, 8h and 24 hours postoperative.

SECONDARY OUTCOMES:
Absolute neutrophil count | The time frame extend from 10 minutes before induction of anesthesia till the first 24 hours postoperative
  Number multiplied by 1000/micro liter,measured before the induction of general anesthesia, 30 min after beginning infusion of the anesthetic agent , then 2h, 8h and 24 hours postoperative.
Total leukocyte count | The time frame extend from 10 minutes before induction of anesthesia till the first 24 hours postoperative
  Number multiplied by 1000/micro liter ,measured before the induction of general anesthesia, 30 min after beginning infusion of the anesthetic agent , then 2h, 8h and 24 hours postoperative.
Neutrophil-lymphocyte ratio (N/L ratio) | The time frame extend from 10 minutes before induction of anesthesia till the first 24 hours postoperative
  measured before the induction of general anesthesia, 30 min after beginning infusion of the anesthetic agent , then 2h, 8h and 24 hours postoperative.
Serum Cortisol level | The time frame extend from 10 minutes before induction of anesthesia till the first 24 hours postoperative
  micro-gram /deciliter by immunoassays techniques.measured before the induction of general anesthesia, 30 min after beginning infusion of the anesthetic agent , then 2h, 8h and 24 hours postoperative.
C-reactive protein serum level | The time frame extend from 10 minutes before induction of anesthesia till the first 24 hours postoperative
  milgram/liter using ELISA technique. measured before the induction of general anesthesia, 30 min after beginning infusion of the anesthetic agent , then 2h, 8h and 24 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Reem Abdelraouf, lecturer, Principal Investigator — Mansoura University